CLINICAL TRIAL: NCT00504426
Title: Dose-ranging Trial of OPC-249 Powder Inhalation in Patients With Pain Due to Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 249-06-002OD
Record Dates: First submitted 2007-07-16; First posted 2007-07-20 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2013-12

CONDITIONS: Pain Due to Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: OPC-249
- 2 (Active Comparator)
  Interventions: Drug: OPC-249
- 3 (Active Comparator)
  Interventions: Drug: OPC-249
- 4 (Active Comparator)
  Interventions: Drug: OPC-249

INTERVENTIONS:
Drug: OPC-249 — 1 pugh/day for 4 weeks (30 IU, 60IU, or 90IU)

SUMMARY:
The purpose of this study is to examine the efficacy and safety of OPC-249 by once daily inhalation at 0 (placebo), 30, 60 or 120 IU for 4 weeks in patients with pain due to osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfill all of the following items

  * Patients with primary osteoporosis
  * Patients who have existing 1-4 vertebral fractures
  * Patients with back pain persisting for one week or more
  * Postmenopausal women between 46 and less than 80 years of age

Ages: 46 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Division of New Product Evaluation and Development
Locations (5):
- Japan (5):
  - Chubu Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo of OPC-249/vial
- OPC-249 (30IU): 30 IU of OPC-249/vial
- OPC-249 (60IU): 60 IU of OPC-249/vial
- OPC-249 (120IU): 120 IU of OPC-249/vial
Period: Overall Study
Arm/Group | Placebo | OPC-249 (30IU) | OPC-249 (60IU) | OPC-249 (120IU)
Started | 32 | 23 | 22 | 24
Completed | 29 | 22 | 18 | 24
Not Completed | 3 | 1 | 4 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | OPC-249 (30IU) | OPC-249 (60IU) | OPC-249 (120IU) | Total
Number analyzed (Participants) | 32 | 23 | 22 | 24 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 2 | 2 | 10
  >=65 years | 28 | 21 | 20 | 22 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (6.0) | 73.0 (5.1) | 73.4 (5.9) | 72.3 (5.9) | 72.6 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 23 | 22 | 24 | 101
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 32 | 23 | 22 | 24 | 101

OUTCOME MEASURES:

1. Primary Outcome: Pain (Subjective Symptom)
Description: Change of pain measured by 100 mm visual analogue scale (VAS) at week4 from baseline.
  Regarding VAS (dotted onto a 100 mm line), 0 mm means "No Pain" and 100 mm means "Worst Pain Imaginable".
Time Frame: Baseline and Week 4
Measure: Mean (Standard Deviation); unit: mm
Groups:
- OPC-249 (30IU): 30 IU of OPC-249 /vial
- OPC-249 (60IU): 60 IU of OPC-249 /vial
- OPC-249 (120IU): 120 IU of OPC-249 /vial
Arm/Group | Placebo | OPC-249 (30IU) | OPC-249 (60IU) | OPC-249 (120IU)
Number analyzed (Participants) | 29 | 22 | 18 | 24
mm | -37.8 (28.7) | -24.5 (27.3) | -40.5 (26.2) | -29.0 (23.7)

2. Secondary Outcome: Improvement Rate of Pain (Doctor's Judgment)
Description: Percentage of participants qualified for improvement of pain by doctor's judgement.
  Qualification: stopped or almost stopped, alleviated, slightly alleviated, unchanged, worsend.
  Improvement defind by "stopped or almost stopped" or "alleviated".
Time Frame: Baseline and Week 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | OPC-249 (30IU) | OPC-249 (60IU) | OPC-249 (120IU)
Number analyzed (Participants) | 29 | 22 | 18 | 24
Percentage of Participants | 69.0 [49.2 to 84.7] | 59.1 [36.4 to 79.3] | 77.8 [52.4 to 93.6] | 66.7 [44.7 to 84.4]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Placebo | OPC-249 (30IU) | OPC-249 (60IU) | OPC-249 (120IU)
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/23 | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 9/32 | 9/23 | 6/22 | 4/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | OPC-249 (30IU) (N=23) | OPC-249 (60IU) (N=22) | OPC-249 (120IU) (N=24)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | OPC-249 (30IU) (N=23) | OPC-249 (60IU) (N=22) | OPC-249 (120IU) (N=24)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Disorder gastrointestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Surfactant protein increase (Investigations) | 3 (3) | 4 (4) | 3 (3) | 1 (1)
Blood pressure rise (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Limbs pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No